CLINICAL TRIAL: NCT00004770
Title: Pilot Compassionate Use Study of Thioctic Acid Treatment in Mitochondrial Myopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Rochester (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11774; URMC-5231
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Mitochondrial Myopathy
Keywords: inborn errors of metabolism; mitochondrial myopathy; rare disease
MeSH Terms: conditions — Mitochondrial Myopathies; Metabolism, Inborn Errors; Rare Diseases | interventions — Thioctic Acid

INTERVENTIONS:
Drug: thioctic acid

SUMMARY:
OBJECTIVES:

I. Assess the efficacy of thioctic acid in treating a single patient with mitochondrial myopathy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: The patient receives one thioctic acid tablet 3 times a day. If patient experiences no side effects after 1 week, 2 tablets are administered and given 3 times a day over 3 months for compassionate use.

The patient is followed at weeks 3, 8, and 12.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Long standing ophthalmoparesis and fatiguable weakness of the limbs
* Mild ataxia and no central nervous system involvement
* History of mitochondrial DNA deletion and a measurable biochemical defect of the respiratory chain
* Steady deterioration in skeletal muscle mass and power over 5 years

--Prior/Concurrent Therapy--

* Previous participation in studies of muscle disease natural history (CRC Protocol 183A)

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Robert Griggs, Study Chair — University of Rochester